CLINICAL TRIAL: NCT05989854
Title: An Individualised 8-week Remote Exercise Intervention to Improve QoL, Cardiometabolic Risk and Physical Activity Level in Men With Prostate Cancer Undergoing ADT Treatment.
Brief Title: The Remote Study: Investigating the Effects or Online Exercise on Quality of Life in Men With Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 956732-956714-101614486
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Exercise; Online; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Exercise arm
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 8 week exercise intervention, 3x/wk

SUMMARY:
Currently, there are few opportunities for patients with cancer to have individual exercise guidance, and this has further been impacted by the Covid-19 pandemic. However, during the pandemic the use of virtual/remote platforms has been crucial in delivering care to cancer patients. The investigators think that remote exercise training may also offer a solution to support positive change in prostate cancer patients. As a result, the investigators have developed a remote/online exercise programme to explore this further.

This study will explore the effectiveness of an 8-week remote exercise and behavioural support intervention, and whether prostate cancer patients feel they benefit from this. The study also aims to see if this sort of exercise programme can be delivered to more prostate cancer patients in the future. This project is open to men with prostate cancer on long term hormone therapy. The intervention will be comprised of one remote supervised session per week, completed 1-1 using an online platform and up to two additional sessions, depending on its suitability for the patient, will be prescribed as unsupervised home-based exercise.

ELIGIBILITY:
Inclusion Criteria:

* Have had an orchiectomy OR;
* Are receiving a GnRH agonist/antagonist OR;
* Are currently receiving Abiraterone, Enzalutamide, Apalutamide or Darolutamide
* Long-term retention is planned (intending to remain on the above stated treatments for at least the next 6 months).

Exclusion Criteria:

* Patients who are currently classed as in active treatment i.e. are currently receiving chemotherapy/radiation therapy (Note: Patients that are included in the study but after inclusion are moved onto chemo/radiation therapy, will still be able to participate in the project).
* Patients who are stratified as high risk for having a cardiovascular event.
* Acute illness; or any musculoskeletal, cardiovascular or neurological disorder that could inhibit or put them at risk from exercising, as determined by screening and their clinician.
* Men with painful or unstable bony metastases.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Prostate | t= 0, 4, 8, 16 & 30 weeks
  Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire. Twenty-seven questions about physical, social/family, emotional and functional well-being are graded from 0-4 (0 = not at all; 4 = very much), yielding a total between 0 and 108.
Functional Assessment of Cancer Therapy | t= 0, 4, 8, 16 & 30 weeks
  Functional Assessment of Cancer Therapy fatigue (FACIT-f) questionnaire. The FACIT-Fatigue is a validated questionnaire that was originally developed for the precise evaluation of fatigue levels in cancer patients with anemia. It consists of 13 questions using a 5 point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). It has been used frequently in the clinical trial setting (please see appendix 1). Responses to each question are added with equal weight to obtain a total score. The range of possible scores is 0-52, with 0 corresponding to the highest level of fatigue and 52 corresponding to the lowest level of fatigue.

SECONDARY OUTCOMES:
Leisure time physical activity | t= 0, 4, 8, 16 & 30 weeks
  Godin Leisure Time Exercise Questionnaire. This is a 3 question self-report questionnaire - indirect measure of physical activity
Physical activity | t= 0, 4, 8, 16 & 30 weeks
  The Dukes Activity Status Index. The Duke Activity Status Index (DASI) is a 12-item questionnaire that utilized self-reported physical work capacity to estimate peak metabolic equivalents (METs).
Cardiovascular risk | t= 0, 4, 8 weeks
  Qrisk3. Estimation of cardiovascular risk based on demographical and physiological parameters
Exercise adherence | weekly for 8 weeks
  Session adherence. The number of sessions attended, and % of scheduled sessions performed. Every exercise session either completed or not completed over the 8 week intervention period
Health status | t= 0, 4, 8, 16 & 30 weeks
  eq-5d-5l. It comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, some problems, severe problems and unable to do. Each level of answer consists of each level of score ranges from 1 to 5. Each participant will have a health status consisting of 5 digits. Using the set of weights from Vietnamese population provided from the EuroGroup, we can convert each EQ-5D health state into a single summary index value. The index value ranges from 0 to 1, higher scores meaning better health quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No de-identified data will be shared with other researchers to protect patient confidentiality